CLINICAL TRIAL: NCT00495950
Title: Prospective Measurement of Post-Treatment Lymphedema in Patients With Melanoma
Brief Title: Prospective Measurement of Post-Treatment Lymphedema
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Clinical Oncology Research Development Program (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2004-0787; 5K12CA088084 (NIH)
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: Melanoma; Lymphedema; Limb Swelling; Questionnaire; Quality of Life; Physical Function; Survey
MeSH Terms: conditions — Melanoma; Lymphedema | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaire
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaires relating to symptoms experienced during and following standard cancer treatment.
  Other Names: Survey

SUMMARY:
The goal of this study is to measure the amount of limb swelling (lymphedema) that sometimes occurs after melanoma treatment, and to find out how people feel and react to the diagnosis and treatment of melanoma.

DETAILED DESCRIPTION:
If you choose to take part in this study, you will have measurements taken of your arms or legs using a Perometer and a bioimpedance machine. The Perometer is a machine that painlessly measures the fluid in your limb using two-directional infrared lights. These lights are located in the frame of the machine that encircles the arm or leg during the measurement. The bioimpedance is a machine that measures the fluid in your arm or leg by passing a very small current through the body similar to an electrocardiogram (EKG). These very small currents are located in electrodes that are placed on the hands and feet during the measurement. Both machines are able to pick up changes in limb size.

You will also be asked to complete a set of questionnaires relating to any symptoms that you may experience in your limbs and/or trunk (chest, stomach, and hip areas) during and following your standard cancer treatment.

Additional questionnaires, along with your limb measurements, will be done at your regularly-scheduled follow-up clinic visits, 3-6 months, 9-12 months, 15-18 months, 21-24 months and 27- 30 months. You will complete the additional questionnaires using a laptop computer or a hardcopy. The measurements and questionnaires will take 45-60 minutes to complete each time.

Some of the data from this study may be sent to the University of Missouri for analysis. The data that is sent will not have any personal identifiers. Researchers at University of Missouri will not be able to link the data to the protected health information or personal identity of any individual participant.

This is an investigational study. Up to 350 patients will take part in this study. All patients will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis (M.D. Anderson pathology) of invasive cutaneous melanoma (stages I-III) will be recruited for participation as they present for their initial clinical evaluation to the University of Texas M.D. Anderson Melanoma and Skin Center.
2. Prior to surgical treatment
3. Patients who can knowledgeably and voluntarily provide an informed consent to participate. The informed consent will be signed and dated.
4. Fluent in English.
5. At least 18 years of age.

Exclusion Criteria:

1. Patients with a prior history of lymphedema or melanoma prior to treatment.
2. Patients who are unable to consent due to other medical illnesses or disorientation to person, place or time.
3. Patients with known distant metastatic disease (Stage IV).
4. Patients with implanted device (pace maker), orthopedic implants, and metal frames.
5. Presence of concurrent malignancy that requires active treatment, such as chemotherapy or biotherapy, prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants with a confirmed diagnosis (M.D. Anderson pathology) of invasive cutaneous melanoma (stages I-III).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2006-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of incidences of lymphedema following surgical treatment of stage I, II, and III cutaneous malignant melanoma | 30 Month Period

CONTACTS AND LOCATIONS:
Overall Officials: Janice N. Cormier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org